CLINICAL TRIAL: NCT04168606
Title: Retrospective Descriptive Study on Retroplacental Hematomas in Finistère
Brief Title: Study on Retroplacental Hematomas in Finistère
Acronym: HEMOPLACENTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0193
Record Dates: First submitted 2019-11-04; First posted 2019-11-19 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Placental Abruption; Placenta Diseases
Keywords: placental abruption
MeSH Terms: conditions — Abruptio Placentae; Placenta Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases with placental abruption: Cases of placental abruption included in our study will be clinically defined and will not be only diagnosed by histological examination.
  All cases will be reviewed by an experienced obstetrician in order to confirm the diagnosis.

SUMMARY:
Cases with placental abruption will be identified by interrogation of two databases of Brest University Hospital between January 2013 and December 2018. First trimester PAPPA and bhCG levels will be recorded. PlGF levels will be measured in women with an available first trimester serum sample. Histological findings in placentas, course of pregnancies, maternal and fetal characteristics will described and compared between cases with and without placental chronic inflammation.

DETAILED DESCRIPTION:
Identification of cases:

Placental abruption cases will be identified by interrogation of two databases of Brest University Hospital between January 2013 and December 2018.

The women diagnosed with placental abruption will be first identified by interrogation of the Medical Registry Department (MRD) of Brest University Hospital and of five other maternities of our county between January 2013 and December 2018, using the keyword "placental abruption".

Simultaneously, placental abruption cases will be identified from the Pathology department files of Brest University Hospital using a computerized database (ADICAP system).

Cases of placental abruption included in the study will be clinically defined and will not be only diagnosed by histological examination. All cases will be reviewed by an experienced obstetrician in order to confirm the diagnosis.

Duplicates, medical termination of pregnancy, marginal abruption, placenta previa, cases without histological examination of the placenta, histological cases without compatible clinical signs and cases from an unselected maternity will be excluded.

Women identified with placental abruption in the period of study will be sent an information letter explaining the study and its purpose. Women who express their opposition to participate to the study will be excluded.

Clinical parameters:

The following data will be recorded from medical files on a computerized database: baseline maternal characteristics including preconceptional Body Mass Index (BMI), tobacco use, drug use (cocaine, cannabis, buprenorphine) medical history (chronic hypertension, chronic nephropathy, diabetes, cardiovascular disease, autoimmune disease, previous venous thromboembolism), blood and rhesus group, obstetrical history, especially past vasculoplacental disorder and past placental abruption, age at delivery. The following pregnancy characteristics will also be collected: method of conception, medication during pregnancy (in particular aspirin and low molecular-weight heparin (LMWH)), gestational diabetes, premature rupture of membrane, pre-eclampsia (according to the American College of Obstetricians and Gynecologists' definition published in 2013, term at pre-eclampsia diagnosis, term at delivery and method of delivery, postpartum complications including postpartum hemorrhage (defined by a blood loss > 500 ml, whatever the mode of delivery), disseminated intravascular coagulation (DIVC), thromboembolic event after delivery and before hospital discharge, intensive care admission and length of stay.

The following fetal characteristics will be recorded: presence and term at diagnosis of intrauterine growth restriction (IUGR), stillbirth, birthweight and sex of the newborn. IUGR will be defined according to the 2013 French College of Obstetricians and Gynecologists guidelines by an estimated fetal weight below the 10th percentile using locally-accepted curve (AUDIPOG) associated with signs of fetal growth pathological restriction.

Placental parameters:

Histopathological examination of the placentas had been performed by two senior perinatal pathologists at Brest University Hospital. Histological findings were recorded by interrogation of the pathology computerized database APIX V7.

Placentas were fixed in 4% buffered formalin. Standard sampling of three blocks in the central area was performed and slides were Hematoxylin, Eosin and Saffron (HES) stained.

Recorded macroscopic findings will correspond to the following items: placenta weight, fetoplacental weight ratio, placental abruption, abnormal placental set-up (only circumvallation), abnormal umbilical cord (villamentous implantation, thin umbilical cord with < 0,8 cm in diameter, presence of a knot), presence and number of placental infarcts, intervillous thrombi and thrombi in a vessel of the chorionic plate affecting ≥ one third of the placental surface.

Recorded microscopic lesions will correspond to the following items according to Amsterdam consensus: maternal vascular malperfusion lesions such as microscopic infarcts, decidual arteriopathy, abnormal villous maturation (hypermature villi or villous agglutination), presence of fetal vascular malperfusion signs such as obliterative fetal vasculopathy or avascular villi, chorangiosis and erythroblastosis, excessive fibrin deposition, chronic inflammation such as villitis or chronic intervillositis of unknown etiology, chronic chorioamniotitis or chronic deciduitis, acute inflammation such as acute villitis, acute chorioamniotitis or funiculitis.

Biological parameters:

First trimester Down syndrome screening results will be collected for each pregnancy.

First trimester pregnancy associated plasma protein-A (PAPP-A) and β-human chorionic gonadotrophin (βhCG) levels had been measured in international unit/liter and converted to multiples of the median (MoM) using the crown-rump length or biparietal diameter measurement when the blood sample was obtained as an estimate of gestational age.

Available blood samples collected at the end of first trimester of pregnancy (between 11 weeks of gestation (WG) and 13+6 WG) for Down syndrome screening stored at -20°C in Biochemistry department of Brest University Hospital will be used for Placental Growth Factor (PlGF) quantification. Measurements will be done with the automated B.R.A.H.M.S KRYPTOR compact PLUS system (B.R.A.H.M.S PlGF plus KRYPTOR: Thermo Fisher Scientific, Hennigsdorf, Berlin) according to the manufacturer's instructions described elsewhere. PlGF levels will be expressed in pg/ml.

Informed written consents were obtained from women whose blood samples had been collected at the end of first trimester.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* who had a placental abruption (clinically defined)
* with an available placental histological examination
* in one of 5 maternities of our county (Finistère, France)
* between January 2013 and December 2018.

Exclusion Criteria:

* Medical termination of pregnancy
* marginal abruption
* placenta previa
* cases without histological examination of the placenta
* histological cases without compatible clinical signs
* cases from an unselected maternity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who had a placental abruption (clinically defined) with an available placental histological examination in one of 5 maternities of our county (Finistère, France) between January 2013 and December 2018.
  Women identified with placental abruption in the period of study will be sent an information letter explaining the study and its purpose. Women who express their opposition to participate to the study will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Histological findings in placentas n°1 | through study completion, an average of one year
  placenta weight
Histological findings in placentas n°2 | through study completion, an average of one year
  presence of an histologic placental abruption
Histological findings in placentas n°3 | through study completion, an average of one year
  presence of an abnormal placental set-up
Histological findings in placentas n°4 | through study completion, an average of one year
  presence of an abnormal umbilical cord
Histological findings in placentas n°5 | through study completion, an average of one year
  presence of thrombi in the chorionic plate or intervillous thrombi
Histological findings in placentas n°6 | through study completion, an average of one year
  presence of maternal vascular malperfusion lesions such as macroscopic or microscopic infarcts, decidual arteriopathy or abnormal villous maturation
Histological findings in placentas n°7 | through study completion, an average of one year
  presence of fetal vascular malperfusion signs such as obliterative fetal vasculopathy or avascular villi
Histological findings in placentas n°8 | through study completion, an average of one year
  presence of chorangiosis or erythroblastosis
Histological findings in placentas n°9 | through study completion, an average of one year
  presence of excessive fibrin deposition
Histological findings in placentas n°10 | through study completion, an average of one year
  presence of chronic inflammation such as villitis or chronic intervillositis of unknown etiology, chronic chorioamniotitis or chronic deciduitis
Histological findings in placentas n°11 | through study completion, an average of one year
  presence of acute inflammation such as acute chorioamniotitis or funiculitis

SECONDARY OUTCOMES:
Maternal first trimester biological markers n°1 | through study completion, an average of one year
  PAPPA
Maternal first trimester biological markers n°2 | through study completion, an average of one year
  Beta HCG
Maternal first trimester biological markers n°3 | through study completion, an average of one year
  PlGF
Course of the pregnancies n°1 | through study completion, an average of one year
  single or twin pregnancy
Course of the pregnancies n°2 | through study completion, an average of one year
  use of aspirin or heparin during pregnancy
Course of the pregnancies n°3 | through study completion, an average of one year
  occurrence of pre-eclampsia
Course of the pregnancies n°4 | through study completion, an average of one year
  occurrence of IUGR
Course of the pregnancies n°5 | through study completion, an average of one year
  occurrence of stillbirth
Course of the pregnancies n°6 | through study completion, an average of one year
  occurrence of premature rupture of membrane
Course of the pregnancies n°7 | through study completion, an average of one year
  occurrence of gestational diabetes
Course of the pregnancies n°8 | through study completion, an average of one year
  term at delivery
Course of the pregnancies n°9 | through study completion, an average of one year
  mode of delivery
Course of the pregnancies n°10 | through study completion, an average of one year
  occurrence of disseminated intravascular coagulation
Course of the pregnancies n°11 | through study completion, an average of one year
  occurrence of postpartum haemorrhage
maternal characteristics n°1 | through study completion, an average of one year
  parity
maternal characteristics n°2 | through study completion, an average of one year
  previous vasculoplacental disorder
maternal characteristics n°3 | through study completion, an average of one year
  BMI before pregnancy
maternal characteristics n°4 | through study completion, an average of one year
  age at delivery
maternal characteristics n°5 | through study completion, an average of one year
  Tobacco use and drug use
maternal characteristics n°6 | through study completion, an average of one year
  chronic hypertension or chronic nephropathy
maternal characteristics n°7 | through study completion, an average of one year
  diabetes
maternal characteristics n°8 | through study completion, an average of one year
  APL syndrome or SLE
maternal characteristics n°9 | through study completion, an average of one year
  previous VTE event
maternal characteristics n°10 | through study completion, an average of one year
  blood group
maternal characteristics n°11 | through study completion, an average of one year
  mode of conception
fetal characteristics n°1 | through study completion, an average of one year
  newborn weight
fetal characteristics n°2 | through study completion, an average of one year
  sex

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest (médecine interne), Brest, France